CLINICAL TRIAL: NCT00260338
Title: Stem Cell Therapy for Vasculogenesis in Patients With Severe Myocardial Ischemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, JKastrup, Professor, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Jens Kastrup
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Myocardial Ischemia; Coronary Heart Disease
Keywords: myocardial ischemia; stem cell; mesenchymal; myocardial perfusion
MeSH Terms: conditions — Myocardial Ischemia; Coronary Disease

ARMS (1):
- Mesenchymal stromal cell (Active Comparator): Mesenchymal stromal cell
  Interventions: Biological: stem cell

INTERVENTIONS:
Biological: stem cell — mesenchymal stromal cell

SUMMARY:
Mesenchymal stem cells from the bone marrow can be stimulated to differentiate into endothelial cells and participate in the development of new blood vessels in ischemic tissue.

The aim of the study is in a phase I/II safety and efficacy study to evaluate the clinical effect of autologous mesenchymal stem cell therapy in patients with severe chronic myocardial ischemia.

DETAILED DESCRIPTION:
Mesenchymal stem cells from the bone marrow can be stimulated to differentiate into endothelial cells and participate in the development of new blood vessels in ischemic tissue.

The aim of the study is in a phase I/II safety and efficacy study to evaluate the clinical effect of autologous mesenchymal stem cell therapy in patients with severe chronic myocardial ischemia.

4o patients with reversible ischemia on a SPECT will be treated with direct intramyocardial injections of autologous isolated and expanded mesenchymal stem cells.Clinical and objective evaluations will be performed at baseline and during 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 80 years Reversible ischemia on a stress SPECT Angina pectoris CCS class >_ 2 Reduced exercise time < 10 min No further revascularization options

Exclusion Criteria:

* Pregnant Present or history of cancer Proliferative retinopathy Systemic severe disease LVEF < 25 % NYHA > II

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Improvement in myocardial perfusion measured by SPECT | 6 months after treatment

SECONDARY OUTCOMES:
Safety | 6 months after treatment
Improvement in myocardial perfusion and function measured by PET and MR | 6 months after treatment
Exercise time | 6 months after treatment
Clinical angina status | 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kastrup, MD DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Cardiovascular Lab. 2014, The Heart Centre, Rigshospitalet, Blegdamcvej 9, Copenhagen, Denmark

REFERENCES:
- [Derived] Mathiasen AB, Haack-Sorensen M, Jorgensen E, Kastrup J. Autotransplantation of mesenchymal stromal cells from bone-marrow to heart in patients with severe stable coronary artery disease and refractory angina--final 3-year follow-up. Int J Cardiol. 2013 Dec 10;170(2):246-51. doi: 10.1016/j.ijcard.2013.10.079. Epub 2013 Oct 28. PMID 24211066